CLINICAL TRIAL: NCT05819216
Title: Partial Body Weight Support Treadmill Training Versus Loaded Treadmill Training in Treatment of Children With Cerebral Palsy: A Randomized Clinical Trial
Brief Title: Support Versus Loaded Treadmill Training in Treatment of Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Abdulmajeed Nasser Alotaibi, Ph.D. candidate, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 45178
Record Dates: First submitted 2023-03-17; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- partial body weight support treadmill training group (Experimental): A set of 24 sessions of partial body weight support treadmill training involve administration of a motorized treadmill with an attached overhead unweighting system of 30% of each participant's body weight will be decreased. The treatment session lasts for 45 min (3 sessions/ week, for 8 weeks).
  Interventions: Device: Treadmill
- loaded treadmill training group (Experimental): A set of 24 sessions of loaded treadmill training includes a motorized treadmill with an additional load (sand bags) attached to the child's lower extremities. A 60% mass lower limb weight will be added.
  Interventions: Device: Treadmill

INTERVENTIONS:
Device: Treadmill — Gait training on treadmill training
  Other Names: Treadmill training

SUMMARY:
Background: Children often suffer from disorders that alter their walking functions, such as cerebral palsy. Task-oriented training is one of the recent interventions to improve gait in children with cerebral palsy (CP). Some studies have shown the effectiveness of Partial Body Weight Support Treadmill Training (PBWSTT) for children with cerebral palsy. Another study supports the effectiveness of Loaded Treadmill Training (LTT) by placing additional weight on the lower extremity. There is still inconsistency in the results of studies advising which weight support or weight addition is more appropriate to use in improving walking in children with cerebral palsy.

Objectives: This study aims to investigate the effectiveness of PBWSTT in the treatment of children with CP. Furthermore, to compare the effectiveness of LTT with PBWSTT.

Methods: Two groups of twenty-two children with spastic cerebral palsy will be involved. Ages 4 to 10 and Gross Motor Functional Classification System (GMFCS) I -III. PBWSTT includes a 45- minute treadmill training session with 30% weight support for group one and LTT by adding 60% weight to lower limb while treadmill training for the second group. Spatiotemporal parameters will be measure additional to balance and endurance functions.

Statistical analysis: Independent t test will be used to detect between group differences and paired t test to detect before and after trial differences. Significance level less than 0.05 and confidence interval 95%.

Study design: Randomized Clinical Trial (Parallel Arm Design).

DETAILED DESCRIPTION:
Study design:

A randomized clinical trial (parallel arm design) will compare the pre- and post-intervention effects of Partial Body Weight Support Treadmill Training and Loaded Treadmill Training.

Participants:

A convenience sampling technique will be used to recruit the children with cerebral palsy aged between 4 and 10 years who had Gross Motor Functional Classification System (GMFCS) from I to III and who could stand and hold. Children will be recruited from the Children's Hospital, Taif, Saudi Arabia.

Interventions:

the pre-and post-intervention effects of Partial Body Weight Support Treadmill Training and Loaded Treadmill Training will be compared. All children will be randomly divided into two groups. Both groups will receive 45-minute treadmill training sessions for 8 weeks (3 sessions per week) with a total of 25 sessions.

First group: (Partial Body Weight Support Treadmill Training) Involve administration of conventional treatment sessions. Further, sessions of Partial Body Weight Support Treadmill Training will be given at the rehabilitation center, outpatient clinic. Partial Body Weight Support Treadmill Training involves a motorized treadmill with an attached unweighting system of 30% of each participant's body weight will be decreased. The treatment session lasts for 45 min (3 sessions/ week, for 8 weeks). A gradual decrease in unweight percentage, that keep knee extended during the stance phase. All procedures will be with assistance and under the observation of a well-trained pediatric physical therapist with an adequate experience with treadmill settings.

Second group: (Loaded Treadmill Training) Will receive a loaded treadmill training in addition to the conventional treatment sessions. Loaded Treadmill Training includes a motorized treadmill with an additional load attached to the child's lower extremities. A 60% mass lower limb weight will be added gradually and upon the child's tolerance. These procedures will be introduced under the supervision of a pediatric physical therapist with experience with treadmill settings. Furthermore, both groups will get the same conventional therapy that includes a range of motion, neurodevelopmental approach, and impairment-based therapies such as stretching and strengthening exercises for 30 minutes three times per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4 to 10.
* Children with CP.
* Diplegic or quadriplegic CP regardless of the tonal abnormality.
* Ambulant with or without assistive devices.
* GMFCS = II-III.
* Able to stand and hold.

Exclusion Criteria:

* Children with hemiplegic CP
* Non-ambulant children
* Children with comorbidities.
* Fixed contractures.
* Severely affected CP.
* Severe cognitive or communicative impairment.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Gait kinematics analysis: 3 dimensional motion capture system | Two time points to measure change over two months. First point, before administration of the first treatment session. Second point immediately after finishing the treatment sessions.
  The system to be employed is the VICON Gait Analysis System, which uses a group of ten cameras to record the motion of the lower limbs.

SECONDARY OUTCOMES:
Gross Motor Functional Measure-66 | Two time points to measure change over two months. First point, before administration of the first treatment session. Second point immediately after finishing the treatment sessions.
  Gross Motor Functional Measure (D and E dimensions) to measure changes in gross motor functions over time. It is an observational instrument used to capture changes in gross motor function in children with cerebral palsy.
Biodex Balance System (BBS) | Two time points to measure change over two months. First point, before administration of the first treatment session. Second point immediately after finishing the treatment sessions.
  IT is a multiaxial device that objectively measures and records an individual's ability to stabilize the involved joint under dynamic stress. It uses a circular platform that is free to move in the anterior-posterior and medial-lateral axes simultaneously.
Biodex System 4 - Isokinetic Dynamometer | Two time points to measure change over two months. First point, before administration of the first treatment session. Second point immediately after finishing the treatment sessions.
  Biodex isokinetic dynamometer allows to evaluate strength, endurance, power and range of motion of all major joints and muscles, and provides highly detailed objective data results of their performance.
Functional Reach Test (FRT) | Two time points to measure change over two months. First point, before administration of the first treatment session. Second point immediately after finishing the treatment sessions.
  It is a single task performance outcome measure that assesses the child's stability to detect the functional dynamic balance, which includes a wooden bar flexible to be adjusted to the child's height.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alaa Ibrahim, PhD, Study Director — Imam Abdulrahman Bin Fisal University
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No